CLINICAL TRIAL: NCT01737294
Title: The Use of QUTENZA™ in Standard Clinical Practice: a Phase IV, Multicentre, European Non-interventional Study
Brief Title: Observation of the Use of QUTENZA™ in Standard Clinical Practice
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: QTZ-EC-0003
Record Dates: First submitted 2012-10-22; First posted 2012-11-29 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Peripheral Neuropathic Pain
Keywords: Phase IV; Peripheral Neuropathic Pain; QUTENZA
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment with QUTENZA: Patients with Peripheral Neuropathic Pain
  Interventions: Drug: Qutenza exposure

INTERVENTIONS:
Drug: Qutenza exposure — Cutaneous patch
  Other Names: Capsaicin

SUMMARY:
This non-interventional study will evaluate the efficacy, tolerability, health related quality of life and use of health resources associated with QUTENZA treatment when QUTENZA is used in standard clinical practice.

The patient's primary diagnosis of peripheral neuropathic pain (PNP) will be classified into subtypes: post-herpetic neuralgia (PHN); HIV-associated neuropathy (HIV-AN); neuropathic back pain; cancer-related neuropathic pain; post-operative & post-traumatic neuropathic pain; and 'other' neuropathies.

DETAILED DESCRIPTION:
A detailed medical history will be taken, with particular emphasis on the primary PNP diagnosis. In addition to all current neuropathic pain medications, all previous therapies (pharmacological and surgical) for PNP from the point of primary diagnosis will be documented.

QUTENZA treatments may be repeated up to every 90 days, in line with the Summary of Product Characteristics document (SPC) as determined by the persistence or return of pain.

Patients who have not required treatment for 365 days or longer may re-enter a treatment cycle if their treating physician decides to retreat them with QUTENZA in the course of standard clinical management.

The duration of participation for each patient will be at least 12 months following first QUTENZA treatment.

Short questionnaires will be completed by the investigator whilst in contact with the patient (either in person or by telephone) at the following time points: 1) Screening prior to the first QUTENZA treatment; 2) at each QUTENZA treatment visit; 3) 2 weeks, 8 weeks following the first QUTENZA treatment 4) 12 weeks following each QUTENZA treatment; 5) any additional contact with the patient outside the protocol schedule.

For patients not returning for retreatment with QUTENZA within any of 6 months, 9 months, and 1 year of their previous QUTENZA treatment further follow-up questionnaires will be completed.

End of study (EoS) is defined as one year after the last patient enrolled receives their first QUTENZA treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. The investigator has decided to treat the patient with QUTENZA as part of provision of standard care for the treatment of peripheral neuropathic pain in non-diabetic adults either alone or in combination with other medicinal products for pain
* 2. The patient is willing and able to comply with protocol requirements for the duration of study participation

Exclusion Criteria:

* 1. The neuropathic painful areas are located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes
* 2. The patient has a history of Type I or Type II diabetes mellitus
* 3. The patient has a diagnosis of any major psychiatric disorder or evidence of cognitive impairment including dementia that, in the opinion of the investigator, may interfere with patient's ability to complete study evaluations
* 4. The patient has received any prior treatment with QUTENZA patches, including blinded patches administered as part of a clinical trial
* 5. The patient has hypersensitivity to capsaicin (i.e. chilli peppers or over-the-counter [OTC] capsaicin products), any QUTENZA excipients or adhesives, or local anesthetics
* 6. The patient has participated in any other clinical study or received an investigational drug within 30 days prior to Screening Visit
* 7. The patient currently engages in any active substance abuse or has a history of chronic substance abuse within 1 year prior to the Screening Visit; or any prior chronic substance abuse (including alcoholism) likely to re-occur during the study period as judged by the investigator
* 8. The patient, in the opinion of the investigator, is not suitable to participate in this NIS for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving QUTENZA for PNP in routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percent change in average pain NPRS (Numeric Pain Rating Scale) scores | From Baseline to mean of all scores recorded between week 2 and week 8 following first treatment
Time to retreatment | Between 1st & 2nd treatments (up to a maximum of 24 months)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)

SECONDARY OUTCOMES:
Proportion of patients achieving 30% decrease in average pain NPRS score | From Baseline to mean of all scores recorded between weeks 2 & 8 following 1st treatment
Proportion of patients achieving 50% decrease in average pain NPRS score | From Baseline to mean of all scores recorded between weeks 2 & 8 following 1st treatment
Percent change in "average pain" NPRS score | From baseline to mean of all scores between Week 2 and Week 8 and Weeks 2 and Week 12 following retreatment(s)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Proportion of patients achieving a 30% decrease in their "average pain" NPRS score (maintenance response) | From Baseline to the mean of all scores between week 2 and week 8 and between week 2 and week 12 following retreatment(s)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Proportion of patients achieving a 50% decrease in their "average pain" NPRS score (maintenance response) | From Baseline to the mean of all scores between week 2 and week 8 and between week 2 and week 12 following retreatment(s)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Absolute change in "average pain" NPRS score | From baseline to the average of pain scores assessed between Weeks 2 & 12 following 1st and subsequent treatment(s)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Proportion of patients achieving a 2-point absolute decrease in their "average pain" NPRS score | From baseline to the average of pain scores assessed between Weeks 2 & 12 following 1st and subsequent treatment(s)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Mean "Average pain" NPRS score | At each time point following 1st and subsequent treatment(s) (up to a maximum of 24 months)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Time (in days) between successive retreatments | Between successive retreatments (up to a maximum of 24 months)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Number of QUTENZA patches used with each treatment | Day 1 of each treatment
Relative change in treatment area size | At first treatment and each retreatment (up to a maximum of 24 months)
  From the 1st treatment to the End of Study (The End of Study is defined as the completion of one year of follow-up from the first Qutenza treatment of the last patient enrolled)
Change in concomitant pain medications | From baseline to End of Study (up to 24 months)
  Percentage remaining on opioids, anticonvulsants, antidepressants
Change in health-related quality of life | From baseline to End of Study (up to 24 months)
  Measured by the EQ-5D (Euroqol-5 dimensions) index
Change in health resource use | From baseline to End of Study (up to 24 months)
  Number of contacts with health professionals in prior 4 weeks
Patient Global Impression of Change | At each follow-up after 1st and subsequent treatment(s) (up to a maximum of 24 months)
  Percentage reporting any degree of improvement. Week 2 after 1st Treatment to End of Study
Patient Self Assessment of Treatment | At 12 weeks, 6 months, 9 months, and 12 months after 1st and subsequent retreatment(s)
  Week 2 after 1st Treatment to End of Study
Change in Work Productivity and Activity Impairment scores | Baseline, week 12, 6 months, 9 months, and 12 months after 1st and subsequent treatment(s)
  Week 2 after 1st Treatment to End of Study
Percentage of patients requiring rescue measures during and after treatment with QUTENZA | From Baseline to End of Study (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Company Medical Expert, Study Director — Astellas Pharma Europe Ltd.
Locations (50):
- Austria (7):
  - Site 103 Abteilung für Anästhesiologie und Intensivmedizin LKH Hartberg, Graz
  - Site 107 Interdisziplinäre Schmerzambulanz Univ. Klinik f. Anästhesiologie und Intensivmedizin Graz, Auenbruggerplatz 29, Graz
  - Site 104 Abteilung für Anästhesie und allgemeine Intensivmedizin Allgemein öffentliches Klinikum-Klagenfurt am Wörthersee St. Veiter Strasse 47, Hartberg
  - Site 105 Abteilung für Anästhesiologie und operative Intensivmedizin Allgemeines Krankenhaus Linz Krankenhausstraße 9, Klagenfurt
  - Site 106 Interdisziplinäre Schmerzambulanz Univ. Klinik f. Anästhesiologie und Intensivmedizin Graz Auenbruggerplatz 29, Linz
  - Site 102 Krankenhaus der Elisabethinen GmbH Abteilung für Anästhesie und Intensivmedizin Elisabethinergasse 14, Vienna
  - Site 101 Krankenhaus der Barmherzigen Brüder Abteilung für Anästhesiologie, Intensivmedizin und Schmerztherapie Johannes von Gott Platz 1, Vienna
- Greece (11):
  - Site 202 Antonios Tavernarakis General Hospital of Athens ''Evangelismos'' - Neurology Clinic, Athens, Attica
  - Site 206 Dimosthenis Mitsikostas Hellenic Navy Hospital of Athens - Neurology Clinic, Athens, Attica
  - Site 205 Antonios Kodounis 251 General Airforce Hospital of Athens - Neurology Clinic, Athens, Attica
  - Site 209 Grigorios Panagopoulos- General Hospital of Athens ''G.Gennimatas'' - Neurology Clinic, Athens, Attica
  - Site 211 Panagiotis Kokotis Aeginitio University Hospital of Athens - A' Neurology Clinic, Athens, Attica
  - Site 208 Alexandros Papadimitriou University General Hospital of Larisa - Neurology Clinic, Larissa, Larisa
  - Site 203 Georgios Georgiadis General Hospital of Thessaloniki ''Ippokratio'' - Neurology Clinic, Thessaloniki, Thessaloniki
  - Site 204 Nikolaos Vlaikidis General Hospital of Thessaloniki ''G.Papanikolaou'' - 3rd Neurology Clinic, Thessaloniki, Thessaloniki
  - Site 213 Mediterraneo Hospital, Athens
  - Site 210 General Hospital of Athens ''G.Gennimatas'' - Neurology Clinic, Athens, Attica
  - Site 212 2 Pindarou and Tseva Str, Koumerki, Thebes
- Italy (7):
  - Site 306 Ospedale regionale "Umberto Parini", Aosta, AO
  - Site 305 Azienda Ospedaliero-Universitaria Consorziale Policlinico, Bari, BA
  - Site 308 Spedali Riuniti di Bergamo, Bergamo, BG
  - Site 301 A.O. Spedali Civili di Brescia, Brescia, BS
  - Site 303 L'INM Neuromed, Istituto Neurologico Mediterraneo, Pozzilli, IS
  - Site 302 Ospedale di Stato della Repubblica di San Marino, Borgo Maggiore, RSM
  - Site 304 Ospedale SS. Annunziata, Taranto, TA
- Portugal (11):
  - Site 608 Hospital Divino Espirito Santo, E.P.E., Açores
  - Site 607 Hospital Garcia da Orta, Almada
  - Site 602 Hospital Professor Dr. Fernando da Fonseca, Amadora
  - Site 603 Hospital Infante D. Pedro EPE, Aveiro
  - Site 611 Centro Hospitalar Cova da Beira - Hospital Universitário Quinta do Alvito, Covilha
  - Site 609 Hospital de Faro, Faro
  - Site 601 Centro Hospitalar Lisboa Norte- Hospital Santa Maria, Lisbon
  - Site 605 Hospital S. João da Madeira, Madeirã
  - Site 606 Centro Hospitalar do Porto-Hospital Santo António, Porto
  - Site 604 Hospital São João, Porto
  - Site 610 Hospital S. Teotónio, Viseu
- Spain (7):
  - Site 702 Hospital Municipal de Badalona, Badalona, Barcelona
  - Site 703 Fundació Puigvert, Barcelona, Barcelona
  - Site 705 Hospital Clinic, Barcelona, Barcelona
  - Site 706 Complejo Hospitalario de Navarra, Pamplona, Pamplona
  - Site 708 Clínica Universitaria de Navarra, Pamplona, Pamplona
  - Site 704 Hospital de Basurto, Bilbao, Vizcaya
  - Site 707 Hospital de Galdakano, Galdakano, Vizcaya
- Switzerland (2):
  - Site 902 Leiter der Schmerzklinik Bethesda-Spital Gellertstrasse 144, Basel
  - Site 901 Schmerzzentrum St. Gallen Kantonspital St.Gallen, Sankt Gallen
- United Kingdom (5):
  - Site 802 West Cumberland General Hospital, Whitehaven, Cumbria
  - Site 804 Royal Infirmary of Edinburgh, Edinburgh
  - Site 803 Western General Hospital, Edinburgh
  - Site 801 Chelsea and Westminster Hospital, London
  - Site 805 Princess Elizabeth Hospital, St Martins

REFERENCES:
- [Derived] Mankowski C, Poole CD, Ernault E, Thomas R, Berni E, Currie CJ, Treadwell C, Calvo JI, Plastira C, Zafeiropoulou E, Odeyemi I. Effectiveness of the capsaicin 8% patch in the management of peripheral neuropathic pain in European clinical practice: the ASCEND study. BMC Neurol. 2017 Apr 21;17(1):80. doi: 10.1186/s12883-017-0836-z. PMID 28431564